CLINICAL TRIAL: NCT05963984
Title: An Open-label, Interventional, Multicenter, Randomized, Phase 2 Study of Fulvestrant With or Without Samuraciclib in Participants With Metastatic or Locally Advanced Hormone Receptor (HR) Positive and Human Epidermal Growth Factor Receptor (HER)2-Negative Breast Cancer (BC)
Brief Title: A Study of Samuraciclib in Combination With Fulvestrant in Metastatic or Locally Advanced Breast Cancer in Adult Participants
Acronym: SUMIT-BC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Carrick Therapeutics Limited (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CT7001_002; 2023-503903-27-00 (Registry Identifier: CTIS); Z0041001 (Other: Pfizer)
Record Dates: First submitted 2023-06-30; First posted 2023-07-27 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Metastatic Breast Cancer; Locally Advanced Breast Cancer; Breast Cancer
Keywords: Metastatic Breast Cancer; Advanced Breast Cancer; Breast Cancer; HR Positive; HER2-Negative
MeSH Terms: conditions — Breast Neoplasms | interventions — Fulvestrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A (Experimental): Participants will receive 360 mg of samuraciclib on cycles of 28 days (Cycle 1 to 6), 56 days (Cycle 7 to 9) and up to 84 days (Cycles 10 onwards in combination with fulvestrant administered monthly, plus an additional dose at Cycle 1 Day 15.
  Interventions: Drug: Samuraciclib; Drug: Fulvestrant
- Arm B (Experimental): Participants will receive 240 mg of samuraciclib on cycles of 28 days (Cycle 1 to 6), 56 days (Cycle 7 to 9) and up to 84 days (Cycles 10 onwards in combination with fulvestrant administered monthly, plus an additional dose at Cycle 1 Day 15.
  Interventions: Drug: Samuraciclib; Drug: Fulvestrant
- Arm C (Experimental): Participants will receive fulvestrant administered monthly, plus additional dose at Cycle 1 Day 15.
  Interventions: Drug: Fulvestrant

INTERVENTIONS:
Drug: Samuraciclib — Samuraciclib tablet by mouth once a day
  Arms: Arm A; Arm B
Drug: Fulvestrant — Injection administered monthly (i.e., every 4 weeks), plus additional dose at Cycle 1 Day 15
  Other Names: Faslodex

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of samuraciclib in combination with fulvestrant versus fulvestrant alone in adult participants with metastatic or locally advanced Hormone Receptor (HR) positive and Human Epidermal Growth Factor Receptor (HER)2-negative breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of ER-positive, HER2-negative locally advanced or metastatic breast cancer.
* Documented objective disease progression while on or within 6 months after the end of the most recent therapy.
* Received prior AI in combination with a CDK4/6i as the last therapy
* Known TP53 mutation status.
* Participants must have measurable disease or bone only disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
* Pre/peri-menopausal participants must have commenced treatment with a luteinizing hormone-releasing hormone (LHRH) agonist at least 4 weeks prior to first dose of study intervention.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤1 with no deterioration over the past 2 weeks.
* Expected life expectancy of >12 weeks in the judgement of the treating investigator.

Exclusion Criteria:

* Inflammatory breast cancer.
* Participants with any other active malignancy within 3 years prior to enrollment, except for adequately treated basal cell or squamous cell skin cancer, or carcinoma in situ of the cervix.
* More than 1 line of endocrine treatment for locally advanced or metastatic disease treatment.
* Inadequate hepatic, renal, and bone marrow function.
* Clinically significant cardiovascular disease.
* Any current or prior central nervous system metastases, carcinomatous meningitis, or leptomeningeal disease.
* Pregnant or breastfeeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-11-16 (Actual); Primary Completion 2025-03-20 (Actual); Study Completion 2025-08-28 (Actual)

PRIMARY OUTCOMES:
Clinical Benefit Response (CBR) | From randomization until Week 24
  CBR is defined as the overall complete response (CR), partial response (PR), or stable disease (SD) ≥ 24 weeks according to RECIST version 1.1 recorded from randomization until disease progression, or death due to any cause.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Time from the date of first dose of study intervention until the first documentation of disease progression, death, withdrawal of consent, or start of new anticancer therapy (assessed up to week 48)
  ORR defined as the proportion of participants who achieved a best overall Response (BOR) of CR or PR per RECIST Version 1.1 from randomization until disease progression, or death due to any cause.
Duration of Response (DOR) | Time from the date of first dose of study intervention until the first documentation of disease progression, death, withdrawal of consent, or start of new anticancer therapy (assessed up to week 48)
  DOR defined as the time from the date of first documentation of objective tumor response (CR or PR) to the earliest documented disease progression per RECIST version 1.1, or death due to any cause.
Progression Free Survival (PFS) | Time from the date of first dose of study intervention until the first documentation of disease progression, death, withdrawal of consent, or start of new anticancer therapy (assessed up to week 48)
  PFS defined as the time from the date of randomization to the earliest documented disease progression per RECIST version 1.1, or death due to any cause.
Incidence and severity of adverse events (AEs) as assessed by the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) v5.0 | From first dose of any study intervention through 28 days after the last dose of any study intervention
  Safety will be assessed by monitoring adverse events and clinically relevant changes in vital signs and clinical laboratory results.
Samuraciclib plasma exposure: Cmax | Day 1 of Cycles 2 and 3 (each cycle is 28 days)
Samuraciclib plasma exposure: Ctrough | Cycle 1 Days 8 and 15; Day 1 of Cycles 2, 3, 4, 5, and 6; and within 28 days of last dose (each cycle is 28 days)
Fulvestrant plasma exposure: Ctrough | Cycle 1 Days 8 and 15; Day 1 of Cycles 2, 3, 4, 5 and 6; and within 28 days of last dose (each cycle is 28 days)

CONTACTS AND LOCATIONS:
Locations (32):
- United States (5):
  - Ocala Oncology Center PL DBA Florida Cancer Affiliates, Ocala, Florida
  - Mfsmc-Hjwci, Baltimore, Maryland
  - Saint Luke's Cancer Institute, Kansas City, Missouri
  - Sidney Kimmel Cancer Center - Jefferson Health, Philadelphia, Pennsylvania
  - The Center for Cancer and Blood Disorders, Fort Worth, Texas
- Hungary (3):
  - Szent Borbala Korhaz, Tatabánya, Komárom-Esztergom
  - Nograd Varmegyei Szent Lazar Korhaz, Salgótarján, Nógrád megye
  - Semmelweis Egyetem, Budapest
- Mexico (6):
  - Actualidad Basada en la Investigación del Cáncer, Guadalajara, Jalisco
  - Renati Innovation S.A.P.I de C.V, Guadalajara, Jalisco
  - Soltmed SMO, Mexico City, Mexico City
  - Cryptex Investigación Clínica S.A. de C.V., Cuauhtémoc
  - Oaxaca Site Management Organization S.C., Oaxaca City
  - Centro de Investigacion Clinica de Oaxaca, Oaxaca City
- Spain (10):
  - Institut Català d'Oncologia - L'Hospitalet, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario Marqués de Valdecilla, Santander, Cantabria Comunidad de
  - Hospital Clinico San Carlos, Madrid, Madrid, Comunidad de
  - Hospital Infanta Cristina, Badajoz
  - Parc de Salut Mar - Hospital del Mar, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - MD Anderson Cancer Center, Madrid
  - Hospital Vithas Málaga, Málaga
  - Hospital Universitario de Salamanca - Complejo Asistencial Universitario de Salamanca, Salamanca
  - Hospital Clinico de Valencia, Valencia
- Turkey (Türkiye) (8):
  - Gulhane Egitim ve Arastirma Hastanesi, Ankara
  - Gazi University, Ankara
  - Dr. Abdurrahman Yurtaslan Ankara Onkoloji Egitim ve Arastırma Hastanesi, Ankara
  - Hacettepe Universite Hastaneleri, Ankara
  - Trakya University, Edirne
  - Istanbul Universitesi Istanbul Tıp Fakultesi Hastanesi, Istanbul
  - TC Saglik Bakanligi Goztepe Prof. Dr. Suleyman Yalcin Sehir Hastanesi, Istanbul
  - I.E.U. Medical Point Hastanesi, Izmir

IPD SHARING:
Plan to Share IPD: No